CLINICAL TRIAL: NCT06014645
Title: The Effect of Different Home Programs on Pain and Mobility Gain After Lumbar Spinal Decompression Surgery
Brief Title: Effectiveness of Home Programs After Lumbar Spinal Decompression Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bursa NRŞ RKÇ
Record Dates: First submitted 2023-08-17; First posted 2023-08-28 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Lumbar Spine Disease
MeSH Terms: conditions — Spinal Diseases | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This program will include reeducation isometric contraction exercises for transversus obdominus, oblique abdominals, multifidus lumborum muscles and strengthening stretching exercises for other extremities. These interventions will be sent to the patients via telerehabitation method and the patients will always have access to the programs and training.
  Interventions: Other: Rehabilitation
- Control Group (Active Comparator): The control group will receive post-operative exercise training and will be encouraged to move as described by Moseley et al., 2004.
  Interventions: Other: Control

INTERVENTIONS:
Other: Rehabilitation — The study group will be given a core stabilization program in addition to education.
  Arms: Intervention Group
Other: Control — The control group will receive post-operative cognitive training and will be encouraged to move.
  Arms: Control Group

SUMMARY:
The study will be conducted with volunteer patients who are followed up by Bursa Çekirge State Hospital Cekirge State Hospital Neurosurgery outpatient clinic and who have undergone lumbar decompression surgery and who meet the study criteria. The cases will be divided into 2 groups by randomization software. The control group will receive post-operative exercise training and will be encouraged to move. The study group will receive a core stabilization program in addition to education via telerehabilitation. The first evaluation will be performed 2 months post-operatively and the second evaluation will be performed 2 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone lumbar decompression surgery without fusion and 2 months of history
* Participate in all necessary follow-up assessments
* Being between 18-65 years old
* Understand simple commands
* Signing the consent form

Exclusion Criteria:

* Presence of a previous spinal fusion surgery
* Presence of malignancy
* Having undergone spine surgery before
* Have any other orthopedic or neurological problem that may affect treatment and assessments
* Situations that prevent communication
* Lack of cooperation during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Baseline VAS at 8 weeks
  On a 10 cm straight line or numeric scale, the patient is asked to mark the pain they feel (0: no pain, 10: excruciating pain).
Tampa Scale for Kinesiophobia (TSK) | Change from Baseline TSK at 8 weeks
  The questionnaire is a 17-item scale developed to measure fear of movement/reinjury. The normal score range is between 17 and 68.
Pain Catastrophising Scale (PCS) | Change from Baseline PCS at 8 weeks
  Scale is used to assess the patient's feelings and thoughts about pain and disaster. The total score ranges from 0 to 52 points. A high score indicates a bad situation.
Roland Morris Disability Questionnaire (RMDQ) | Change from Baseline RMDQ at 8 weeks
  The RMDQ is a self-administered questionnaire consisting of 24 items reflecting various activities of daily living. Each item is scored 1 if it is declared applicable to the participant and 0 otherwise, so that the total score can range from 0 (no disability) to 24 (severe disability).
Lumbar region flexibility in flexion extension lateral flexion directions | Change from Baseline flexibilty tests at 8 weeks
  The subject stands on a block and then performs lumlal flexion with knees straight. The distance above the block with the finger is recorded with a negative sign and the distance below the block is recorded with a positive sign. The subject stands in front of a wall. The pelvis and trunk should be in contact with the wall. The subject is asked to perform lumbar extension. The distance between the sternal notch and the wall is measured and noted. The subject stands in front of a wall with hands next to the trunk. The subject is asked to perform lumbar lateral flexion. The distance from the first position to the last position is measured using the middle finger as a base and noted.
Lumbar region endurance flexor and extensor | Change from Baseline endurance tests at 8 weeks
  The participant is placed prone on a treatment bed with the upper edge of the iliac crests flush with the edge of the bed. The lower body is secured to the bed with two straps. At the beginning of the test, participants cross their arms over their chest and remain in a neutral position for as long as possible. The time the position can be maintained is measured using a stopwatch. Participants are held in a supine position with both hips and knees flexed 90 degrees and the trunk flexed 60 degrees on a wedge. Stabilization is achieved with support from the back of the foot. After the wedge is moved back 10 cm, the participants maintain their body position for as long as possible. The time from the moment the wedge is moved back to the moment the participant re-establishes contact with the wedge is measured.
Functional Reach Test (FRT) | Change from Baseline FRT at 8 weeks
  The subject stands sideways next to a wall and flexes the shoulder 90 degrees. The 3rd metacarpal level is marked on the wall. The subject reaches as far as he/she can without taking a step. The 3rd metacarpal line is marked again. The difference between the marks is measured and noted.
Stair Climbing Test (SCT) | Change from Baseline SCT at 8 weeks
  The time (in seconds) taken to ascend and descend one flight of stairs is noted. A 9-step ladder with a 20 cm step height and a handrail is used. You are instructed to ascend and descend the stairs as quickly but safely as possible. The use of a handrail and walking aid is allowed if necessary. Timing starts with the start signal and ends when the participant has lowered both feet to ground level. The participant can stop and rest if necessary, but the timing continues.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, PhD, Study Director — Muğla Sıtkı Koçman University; Mustafa Yalçın, MSc, Principal Investigator — Bursa Çekirge State Hospital; Baki Umut Tuğay, PhD, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Bursa Çekirge State Hospital, Bursa, Osmangazi, Turkey (Türkiye)